CLINICAL TRIAL: NCT06241625
Title: Virtual Reality (VR) Based Vision Test in Subjects With Age-related Macular Degeneration (AMD)
Brief Title: Virtual Reality Based Vision Test in Patients With AMD
Acronym: GA-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augenklinik Zurich West (Other)
Collaborators: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APL-GA-001
Record Dates: First submitted 2023-01-05; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-Visual Function Test (Experimental): Assessment of virtual reality based vision function in Patients with AMD
  Interventions: Diagnostic Test: Virtual Reality (VR) Contrast Function Test

INTERVENTIONS:
Diagnostic Test: Virtual Reality (VR) Contrast Function Test — Patients perform a new Virtual Reality (VR) Contrast Function Test

SUMMARY:
To assess the usability, tolerability, and repeatability of the set of VR headset-based tasks.

DETAILED DESCRIPTION:
In order to bridge the gap between the existing functional measures and AMD lesions, researchers are considering the use of VR tools.

This study is designed to assess the contrast sensitivity function mapping test (CSF radial sweep) in an elderly population with AMD.

The primary objective of this study is to assess the usability, tolerability, and repeatability of the set of VR headset-based tasks.

The secondary objective of this study is to assess the relationship between the metrics generated by VR-based functional tasks and the metrics derived from conventional clinical measurements of retinal anatomy and visual function.

The primary efficacy endpoint is the Contrast sensitivity function (CSF) area under curve (AUC) correlation to Snellen BCVA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age diagnosed with AMD
2. Subject Snellen BCVA score is 20/100 or better
3. Ability to undergo quality optical coherence tomography (OCT) imaging
4. Willing and able to give written informed consent

Exclusion Criteria:

1. Unwilling to use headset
2. Previous negative experience with a VR headset (eg, motion sickness, discomfort)
3. Any known oculomotor impairment that would impact the ability of the subject to perform the tasks (eg, nystagmus, proptosis, apraxia of eyelid opening)
4. Any manifest neurological or cognitive condition that would impair the subject's understanding or performance on the test (eg, Alzheimer's disease, Parkinson's disease)
5. Any physical limitations that would prohibit the use of the VR headset (eg, neck problems)

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Usability, tolerability and repeatability | 20 minutes
  The primary objective of this study is to assess the usability, tolerability, and repeatability of the set of VR headset-based tasks. To assess the usability and tolerability a patient survey is performed.

SECONDARY OUTCOMES:
Contrast sensitivity function (CSF) | 10 minutes
  Contrast sensitivity function (CSF) in decibel as area under curve (AUC). The CSF is also correlated to Snellen best corrected visual acuity (BCVA)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Michels, MD, Principal Investigator — Augenklinik Zurich West
Locations (1):
- Augenklinik Zurich West, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No